CLINICAL TRIAL: NCT02846844
Title: Study Patients With Chemotherapy-induced Polyneuropathy Are Randomized for an Integrated Program (IP) Including Massage, Mobilization in Posture and Transport Layers, Physical Exercises or With Whole-body Vibration Platform Training
Brief Title: Patients With Chemotherapy-induced Polyneuropathy Are Treated With an Integrated Program Including Massage, Mobilization in Posture and Transport Layers, Physical Exercises or With Whole-body Vibration Platform Training
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard Schlenk, Prof. Dr., University of Ulm
Other Study IDs: PI-PNP - _01_10
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Polyneuropathy
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: * Whole body vibration training
  * manuelle therapy
  * exercises for power and coordination
  * performance training as needed
- Group B: * manuelle therapy
  * Exercises for power and coordination
  * Performance training as needed

SUMMARY:
In a Phase-III Study Patients With Chemotherapy-induced Polyneuropathy (NCI CTC Grade 2/3) Are Randomized for an Integrated Program (IP) Including Massage, Mobilization in Posture and Transport Layers, Physical Exercises (Standard) or With Whole-body Vibration (WBV) Platform Training (Experimental).

DETAILED DESCRIPTION:
Subjects with a haematological malignancy or solid and a diagnosis of a chemotherapy-induced polyneuropathy. In a phase-III study patients with chemotherapy-induced polyneuropathy (NCI CTC grade 2/3) are randomized for an integrated program (IP) including massage, mobilization in posture and transport layers, physical exercises (standard) or with whole-body vibration (WBV) platform training (experimental). 15 training sessions in a time period of 12 to 15 weeks were intended. Evaluation included locomotor and neurological tests and self-assessment-tools. The primary objective of the study was the physical fitness and coordination assessed by the chair-rising test (CRT).

ELIGIBILITY:
Inclusion Criteria:

Patients 18 to 70 years of age with solid and hematological neoplasms suffering from chemotherapy-induced polyneuropathy grade II-III according to National Cancer Institute Common Toxicity Criteria (NCI CTC, version 3.0) and pathological chair-rising test (CRT)28 ( ≥10 s) were eligible

Exclusion Criteria:

* psychiatric disorders
* plasmatic coagulation disorders
* thrombotic/thromboembolic events within 6 months before randomization
* severe neurological disorders like seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a haematological malinancy or solid and a diagnosis of a chemotherapy-induced polyneuropathy.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2010-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
• The primary endpoint of the study was achievement of normal values (<10 seconds) in the chair-rising test at the last assessment 4 weeks after the last intervention. | 12 weeks

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Schonsteiner SS, Bauder Missbach H, Benner A, Mack S, Hamel T, Orth M, Landwehrmeyer B, Sussmuth SD, Geitner C, Mayer-Steinacker R, Riester A, Prokein A, Erhardt E, Kunecki J, Eisenschink AM, Rawer R, Dohner H, Kirchner E, Schlenk RF. A randomized exploratory phase 2 study in patients with chemotherapy-related peripheral neuropathy evaluating whole-body vibration training as adjunct to an integrated program including massage, passive mobilization and physical exercises. Exp Hematol Oncol. 2017 Feb 7;6:5. doi: 10.1186/s40164-017-0065-6. eCollection 2017. PMID 28194306